CLINICAL TRIAL: NCT07370519
Title: Safety and Efficacy of Lactobacillus Reuteri for Androgenetic Alopecia: A Single-Center, Randomized, Double-Blind, Placebo-Controlled Trial
Brief Title: Topical Application of Lactobacillus Reuteri for Androgenetic Alopecia
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Shenzhen People's Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: LL-KY-2025109-02
Record Dates: First submitted 2026-01-17; First posted 2026-01-27 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2025-12

CONDITIONS: Androgenetic Alopecia (AGA)
Keywords: Androgenetic Alopecia; Lactobacillus reuteri
MeSH Terms: conditions — Alopecia | interventions — Minoxidil; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Test Group (Experimental): Daily application of 1 sachet containing Lactobacillus reuteri powder (≈10^9 CFU) dissolved in 1 mL normal saline within a brown glass vial. After thorough mixing, 1 mL of the probiotic solution was topically applied to the scalp using cotton swabs following scalp cleansing. Participants refrained from hair washing for ≥6 hours post-application. Applied once daily for 12 months.
  Interventions: Biological: Lactobacillus reuteri
- Inactivated Control Group (Other): Daily application of 1 sachet containing inactivated Lactobacillus reuteri powder (≈10^9 CFU pre-inactivation) dissolved in 1 mL normal saline within a brown glass vial. After thorough mixing, 1 mL of the solution was topically applied to the scalp using cotton swabs following scalp cleansing. Participants refrained from hair washing for ≥6 hours post-application. Applied once daily for 12 months.
  Interventions: Biological: Inactivated Lactobacillus reuteri
- Positive Control Group (Active Comparator): Commercially available 5% minoxidil tincture was aliquoted into brown glass vials (1 mL/vial). Following daily scalp cleansing, 1 mL solution was topically applied to the scalp. Participants refrained from hair washing for ≥6 hours post-application. Applied once daily for 12 months.
  Interventions: Drug: 5% Minoxidil
- Negative Control Group (Placebo Comparator): Normal saline was aliquoted into brown glass vials (1 mL/vial). Following daily scalp cleansing, 1 mL solution was topically applied to the scalp using cotton swabs. Participants refrained from hair washing for ≥6 hours post-application. Applied once daily for 12 months.
  Interventions: Drug: Normal Saline

INTERVENTIONS:
Biological: Lactobacillus reuteri — Daily application of 1 sachet containing Lactobacillus reuteri powder (≈10^9 CFU) dissolved in 1 mL normal saline within a brown glass vial. After thorough mixing, 1 mL of the probiotic solution was topically applied to the scalp using cotton swabs following scalp cleansing. Participants refrained from hair washing for ≥6 hours post-application. Applied once daily for 12 months.
  Arms: Test Group
Biological: Inactivated Lactobacillus reuteri — Daily application of 1 sachet containing inactivated Lactobacillus reuteri powder (≈10^9 CFU pre-inactivation) dissolved in 1 mL normal saline within a brown glass vial. After thorough mixing, 1 mL of the solution was topically applied to the scalp using cotton swabs following scalp cleansing. Participants refrained from hair washing for ≥6 hours post-application. Applied once daily for 12 months.
  Arms: Inactivated Control Group
Drug: 5% Minoxidil — Commercially available 5% minoxidil was aliquoted into brown glass vials (1 mL/vial). Following daily scalp cleansing, 1 mL solution was topically applied to the scalp. Participants refrained from hair washing for ≥6 hours post-application. Applied once daily for 12 months.
  Arms: Positive Control Group
Drug: Normal Saline — Normal saline was aliquoted into brown glass vials (1 mL/vial). Following daily scalp cleansing, 1 mL solution was topically applied to the scalp using cotton swabs. Participants refrained from hair washing for ≥6 hours post-application. Applied once daily for 12 months.
  Arms: Negative Control Group

SUMMARY:
This is a single-center, randomized, double-blind, placebo-controlled clinical trial designed to evaluate whether topical application of Lactobacillus reuteri can safely and effectively treat androgenetic alopecia. The study is based on the concept that balancing the scalp's microbial community may support hair follicle function. Participants will be randomly assigned to one of four groups receiving either active probiotic solution, inactivated probiotic solution (control for non-viable bacterial effects), a saline placebo, or the standard treatment 5% minoxidil solution for 12 months. Neither participants nor assessing clinicians will know the assigned treatment. The main goal is to measure improvement in hair count per square centimeter after one year. Additional measures include changes in hair thickness and quality. This research seeks to provide high-quality scientific evidence on a new microbiome-targeting approach, offering future patients and healthcare providers insights into a potential alternative or complementary treatment strategy for hair loss.

ELIGIBILITY:
Inclusion Criteria:

1. Patients meeting AGA diagnostic criteria (confirmed by medical history, clinical presentation, and trichoscopy) classified as Norwood-Hamilton stage II-IV or Ludwig grade I-III;
2. Provision of informed consent and voluntary participation;
3. Aged 18-60 years with generally good health status;
4. No use of any hair loss medications within the past six months;
5. Absence of alopecia areata, local infections, or neuromuscular disorders.

Exclusion Criteria:

1. AGA progression >5 years;
2. Active skin disease (e.g., psoriasis flare) or uncontrolled diabetes/CVD;
3. Investigator-assessed protocol non-feasibility.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 388 (Estimated)
Dates: Start 2026-01-25 (Estimated); Primary Completion 2027-01 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Hair Density | The follow-up periods are set at 1, 3, 6, and 12 months after the initial treatment
  Hair density is quantified by counting all visible growing hairs in a unit area of the scalp using a trichoscope

SECONDARY OUTCOMES:
Hair Diameter | The follow-up periods are set at 1, 3, 6, and 12 months after the initial treatment
  Trichoscopy is used to measure the average hair shaft diameter (cross-sectional thickness) of all growing hairs in a defined scalp area.

CONTACTS AND LOCATIONS:
Locations (1):
- Shenzhen People's Hospital, Shenzhen, Guangdong, China

IPD SHARING:
Plan to Share IPD: No